CLINICAL TRIAL: NCT04206683
Title: How Does Cerebral-measured Oxygenation and Burst Suppression Correlate Cranially Frontally in Children Between 6 and 36 Months Old, During General Anesthesia and Open Thoracic Surgery Supported by Cardiac Pulmonary Machine
Brief Title: Cerebral Oxygenation and Burst Suppression
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 1066-18 20181230
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Coronary Syndrome; Pediatric
Keywords: brain saturation; burst suppression; general anesthesia; pediatric
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
investigators want to observe a group of pediatric patients who are going to undergo open thoracic surgery at Queen Silvia's child and youth hospital, Sahlgrenska University Hospital. Population that has been selected is between 6-36 months due to the fact that the physiological development does not differ significantly with respect to drug response and circulation. During general anesthesia and surgery, investigators will use an NIRS). A sensor is placed frontally on the head.

This comparative study will study the relationship between regional oxygenation frontal and 2/4-channel EEG. An EEG sensor with adhesive will also be attached to the frontal on patient's forehead next to tendons from NIRS.

Participants will be consulted consecutively at the thoracic surgeon who will undergo open thoracic surgery with the support of the hair removal machine and who have the intended age for the study at Queen Silvia's Children's and Youth Hospital, Salhgrenska University Hospital.

Peroperatively, data collection will occur in 5-minute intervals for frontal and occipital measurements. The measurements are started before the patient is anesthetized and terminated when the patient is awakened.

Usual monitoring parameters under general anesthesia will be collected and documented, see protocol.

DETAILED DESCRIPTION:
Children who are routinely operated for surgery that cause high levels of circulatory changes (e.g., heart surgery) are currently routinely used to monitor the so-called regional oxygenation technique over the brain, (NIRS). Near infrared spectroscopy (NIRS) is a technique for measuring regional oxygen saturation, indirectly autoregulation in the brain. NIRS use has clinically resulted in an increased possibility of detecting episodes of regional ischemia that had not previously been recognized. Investigators do not know for sure what these episodes of impaired oxygenation in the brain can mean if not detect them in time and thus can correct them. There is no such research that has studied it in children. Investigators know that impaired oxygenation in the brain can occur with severe immediate blood loss. Investigators in the research group have been able to observe that in children who are otherwise healthy and who are operated for cranioplasty procedures <1 year old, when they have ongoing heavy bleeding, the oxygenation in the brain and sometimes sharply decreases before investigators can replace the blood loss, even though the blood pressure can be maintained adequately . Peroperative hypovolaemia is a factor that risks disrupting autoregulation in the brain. Regarding which median arterial pressure (MAP) is required to maintain intact autoregulation under general anesthesia, a scientific consensus is still lacking. Dagal & Lam have shown that an MAP between 50-150 mmhg in adults indicates intact autoregulation, even though they claim that there is great individual variation. Research relating to children and autoregulation is limited, however, there is research on middle arterial pressure (MAP). Today at Drottning silvia's children and youth hospital -thorax surgeon, the Sahlgrenska University Hospital uses a monitor whose brand is called INVOS and which uses NIRS technology.

NIRS e.g. works practically by attaching a sensor to the skin in the area where monitoring is to be performed. By illuminating skin and underlying tissue with infrared light in spectra 700 to 1100 nm, it is possible to measure regional oxygen saturation in different tissues. In cerebral measurement, the sensor is placed frontally, just down the hairline. NIRS then returns absolute values (0-100%) of cerebral oxygen saturation frontally in the area where the sensor is located.

Today, NIRS is routinely used during open-hearth surgery. NIRS may indicate when ischemia or ongoing impaired autoregulation occurs. However, the weakness of the technique may be that even when a circulating organ does not extract oxygen, the NIRS value is high, which means that investigators cannot be completely sure of the values when they are high if other parts that affect the value (pH, mean arterial pressure etc.) are affected negatively. This means that supplementation with EEG e.g. BIS or Masimo technology could increase the possibility that even when "false for high values of NIRS" are detected and thus treatable. Regarding EEG and use on children, studies on deep anesthesia and burst suppression, where in their method similar technical equipment of BIS was used, which intenser in this study to detect burst suppression. Otherwise, the BIS or Masimo technique is used clinically during child anesthesia to part also, for example, at so-called. procedure investigations when one wants rapid flow rates of the study for a certain time, but also in the monitoring of children who have ongoing epileptic seizures when the technique has shown that it detects burst suppression. This new area of studying BS and utilizing and possibly this technology during open heart surgery, if possible, could increase safety even more for these many times already vulnerable children. Investigators want to observe a group of pediatric patients who will undergo open thoracic surgery with the support of a heart lung machine at Drottning Silvia's child and youth hospital, Sahlgrenska University Hospital. The purpose of the study is to study how the regional oxygenation one of the brain possibly has an influence on the emergence of so-called burst suppression. Population that has been selected is between 6-36 months due to the fact that the physiological development does not differ significantly with respect to drug response and circulation. Investigators intend to study 15 children according to statistical calculation see below. The time for data collection of the study is estimated at approx. 12 months.

ELIGIBILITY:
Inclusion Criteria:

* children between 6-36months

Exclusion Criteria:

* brain diseases

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This comparative study will study the relationship between regional oxygenation frontal and 2/4-channel EEG). An EEG sensor with adhesive will also be attached to the frontal on patient's forehead next to tendons from NIRS.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
burst suppression (BS). Time of BS-percent during 1 minute, using Bispectral index monitor | 1 minute
  percent 0-100 higher value worse
regional cerebral saturation, NIRS method will be used | 1 minute
  percent 0-100 high value good

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg, Children Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No